CLINICAL TRIAL: NCT05299983
Title: MsFLASH: Living a Healthy Menopause, Aim 2 Randomized Controlled Trial of MyMenoPlan
Brief Title: MyMenoPlan: Online Resource for Improving Women's Menopause Knowledge and Informed Decision-making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Andrea Z. LaCroix, PhD, Distinguished Professor of Epidemiology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 140604
Record Dates: First submitted 2022-03-01; First posted 2022-03-29 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Menopause; Premenopause; Postmenopause
Keywords: Computer-Assisted Decision Making; Internet-Based Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyMenoPlan (Experimental): Participants are asked to spend at least 20 minutes on the website (MyMenoPlan) assigned to them.
  Interventions: Other: MyMenoPlan
- Control (Active Comparator): Participants are asked to spend at least 20 minutes on at least one of the following websites or other websites of their choice:
  1. North American Menopause Society: https://www.menopause.org/for-women
  2. National Institute on Aging: https://www.nia.nih.gov/health/topics/menopause
  3. The Office on Women's Health-Menopause: https://www.womenshealth.gov/menopause
  Interventions: Other: Control

INTERVENTIONS:
Other: MyMenoPlan — Participants are asked to spend at least 20 minutes on the website (MyMenoPlan) assigned to them.
  Arms: MyMenoPlan
Other: Control — Participants are asked to spend at least 20 minutes on at least one of the following websites:
  1. North American Menopause Society: https://www.menopause.org/for-women
  2. National Institute on Aging: https://www.nia.nih.gov/health/topics/menopause
  3. The Office on Women's Health-Menopause: https://www.womenshealth.gov/menopause
  Arms: Control

SUMMARY:
As part of a National Institute on Aging -funded R01, the investigators developed an evidence-based, multi-media digital resource entitled MyMenoPlan to help women learn about the menopause transition, and the symptoms and treatments of perimenopause/menopause. MyMenoPlan is also designed to help women learn about the effectiveness of treatments for a comprehensive list of midlife symptoms and compare treatments that may help with the specific symptoms women are experiencing.

DETAILED DESCRIPTION:
The purpose of this research study is to:

1. Investigate how women randomly assigned to visit MyMenoPlan use the website (time spent on website, treatment and symptom page views, use of interactive tools, and use of the MyMenoPlan tool).
2. Compare the ratings of women randomly assigned to MyMenoPlan to those randomly assigned to other menopause websites for perceived quality of information, readability, self-efficacy, and credibility of these online menopause resources.

ELIGIBILITY:
Inclusion Criteria:

* As stated above

Exclusion Criteria:

* N/A

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on self-representation of gender identity this study includes females, non-binary people and transgender men defined as follows:
  Non-binary: a non-binary person is someone who does not identify as exclusively a man or a woman.
  Transgender male: A transgender male is a man who was assigned female at birth.
Enrollment: 410 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Z. LaCroix, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Snyder LB, Newton KM, Ng HX, Reed SD, Guthrie KA, Zambrano V, LaCroix AZ. Positive impact of a menopause website - MyMenoplan.org - on treatment intentions, knowledge, and decision making: A randomized controlled trial. Maturitas. 2025 Aug;199:108630. doi: 10.1016/j.maturitas.2025.108630. Epub 2025 Jun 5. PMID 40505527

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligibility screening and quality control checks resulted in exclusion of 503. Internet recruited studies requires careful quality control checks for fraudulent participants.
Groups:
- Control: Participants are asked to spend at least 20 minutes on at least one of the following websites or other websites of their choice:
  1. North American Menopause Society: https://www.menopause.org/for-women
  2. National Institute on Aging: https://www.nia.nih.gov/health/topics/menopause
  3. The Office on Women's Health-Menopause: https://www.womenshealth.gov/menopause
  Control: Participants are asked to spend at least 20 minutes on at least one of the following websites:
  1. North American Menopause Society: https://www.menopause.org/for-women
  2. National Institute on Aging: https://www.nia.nih.gov/health/topics/menopause
  3. The Office on Women's Health-Menopause: https://www.womenshealth.gov/menopause
Period: Overall Study
Arm/Group | MyMenoPlan | Control
Started | 200 | 210
Completed | 200 | 210
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MyMenoPlan | Control | Total
Number analyzed (Participants) | 200 | 210 | 410
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (4.0) | 49.4 (3.8) | 49.3 (3.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 210 | 410
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 9 | 8 | 17
  White | 153 | 154 | 307
  Black | 18 | 28 | 46
  Asian | 2 | 6 | 8
  Native American, Native Hawaiian, Pacific Islander | 3 | 3 | 6
  Multiethnic | 12 | 9 | 21
  Other | 2 | 2 | 4
  Unknown/not reported | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  High school or less | 23 | 42 | 65
  Some college or vocational training | 81 | 87 | 168
  College graduate | 46 | 42 | 88
  Post-graduate degree | 50 | 37 | 87
  Unknown | 0 | 2 | 2
Education (years) [Mean (Standard Deviation); unit: years] | 15.2 (2.3) | 14.7 (2.3) | 14.96 (2.29)
Difficulty paying for basics [Count of Participants; unit: Participants]
  A lot | 30 | 31 | 61
  Some | 63 | 83 | 146
  None | 105 | 93 | 198
  Unknown | 2 | 3 | 5
Menopause Stage [Count of Participants; unit: Participants]
  Premenopause | 18 | 23 | 41
  Perimenopause | 109 | 102 | 211
  Postmenopause | 54 | 66 | 120
  Don't know - IUD | 9 | 10 | 19
  Don't know - hysterectomy but kept ovaries | 8 | 9 | 17
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Perceived Quality of Information
Description: This 7-item, 5-point Likert scale (1- Strongly disagree to 5 - Strongly agree) is adapted from the Post-Study System Usability Questionnaire (PSSUQ) in Lewis (1995). The range of this scale is 1-5. The items in this scale were averaged with a higher score meaning higher on this outcome (perceived quality of information).
  Items:
  1. Reading the information made me feel in more control of my perimenopause/menopause.
  2. The information on the website(s) was helpful to me.
  3. I found the information I was looking for.
  4. The information answered my questions about perimenopause/menopause.
  5. I liked the website (s).
  6. I would have liked more in-depth information. (reverse-coded)
  7. The website(s) were fairly comprehensive about perimenopause /menopause.
Time Frame: Each survey question is answered after spending at least 20 minutes on the assigned website(s)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyMenoPlan | Control
Number analyzed (Participants) | 200 | 210
score on a scale | 4.1 (0.59) | 3.7 (0.73)
Statistical Analysis 1: Comparison: MyMenoPlan vs Control; Test type: Superiority; p < .001, Chi-squared

2. Primary Outcome: Readability
Description: This 2-item, 5-point Likert (1- Strongly disagree to 5 - Strongly agree)scale was derived from the Standardized User Experience Percentile Rank Questionnaire (SUPR-Q) in Sauro (1995). The range of this scale is 1-5. The items in this scale were averaged with a higher score meaning higher on this outcome (readability).
  Items:
  1. The information I read was clear.
  2. The information I read was easy for me to understand.
Time Frame: Each survey question is answered after spending at least 20 minutes on the assigned website(s)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyMenoPlan | Control
Number analyzed (Participants) | 200 | 210
score on a scale | 4.6 (0.52) | 4.4 (0.67)
Statistical Analysis 1: Comparison: MyMenoPlan vs Control; Test type: Superiority; p = 0.02, Chi-squared

3. Primary Outcome: Self-Efficacy for Managing Menopause Symptoms
Description: This is a newly developed Likert scale (1- Strongly disagree to 5 - Strongly agree) for assessing participants' beliefs in their own abilities in managing menopausal symptoms. The range of this scale is 1-5. The items in this scale were averaged with a higher score meaning higher on this outcome (self-efficacy).
  Items:
  1. If I want to, I am certain I could figure out the treatments or coping strategies that would work best for me.
  2. I feel I could treat or cope with my symptoms of perimenopause/menopause if I want to.
Time Frame: Each survey question is answered after spending at least 20 minutes on the assigned website(s)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyMenoPlan | Control
Number analyzed (Participants) | 200 | 210
score on a scale | 4.0 (0.66) | 3.9 (0.71)
Statistical Analysis 1: Comparison: MyMenoPlan vs Control; Test type: Superiority; p = 0.22, Chi-squared

4. Primary Outcome: Credibility
Description: This 2-item, 5-point Likert (1- Strongly disagree to 5 - Strongly agree) scale was derived from the Standardized User Experience Percentile Rank Questionnaire (SUPR-Q) in Sauro (1995). The range of this scale is 1-5. The items in this scale were averaged with a higher score meaning higher on this outcome (credibility).
  Items:
  1. The information is credible.
  2. The information is trustworthy.
Time Frame: Each survey question is answered after spending at least 20 minutes on the assigned website(s)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyMenoPlan | Control
Number analyzed (Participants) | 200 | 210
score on a scale | 4.3 (0.66) | 4.4 (0.65)
Statistical Analysis 1: Comparison: MyMenoPlan vs Control; Test type: Superiority; p = 0.45, Chi-squared

ADVERSE EVENTS:
Time Frame: Participants were asked to spend at least 20 minutes reviewing websites.
Arm/Group | MyMenoPlan | Control
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/210
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/210
Other Adverse Events (participants affected / at risk) | 0/200 | 0/210

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT05299983/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT05299983/SAP_001.pdf
  • Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT05299983/ICF_002.pdf